CLINICAL TRIAL: NCT03268434
Title: Evaluation of Metacognitive Training for Depression (D-MCT) in Outpatient Psychiatric-psychotherapeutic Care: Randomized Controlled Trial
Brief Title: Evaluation of Metacognitive Training for Depression (D-MCT) in Outpatient Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Asklepios Kliniken Hamburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LJ05207
Record Dates: First submitted 2017-08-03; First posted 2017-08-31 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Unipolar Depression
Keywords: Depression; Metacognition; CBT; D-MCT; cognitive bias
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double Blind (Investigator, Outcome Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-MCT Group (Experimental): Metacognitive Training for Depression (D-MCT), 8 sessions (60min); once a week over a period of 8 weeks. Metacognitive Training for depression (D-MCT) is a low-threshold, easy to administer group intervention. It aims at the reduction of depressive symptoms by changing cognitive biases; not only biases targeted in cognitive behavioral therapy but also those identified by basic research.
  Interventions: Behavioral: D-MCT
- Cognitive remediation (Active Comparator): A computerized cognitive remediation program that covers several cognitive domains, such as attention, visuomotor skills, and Memory.The difficulty level adapts automatically to the performance level of each patient. At the end of each session, the patient receives individual feedback on his or her performance.; 8 sessions (60min), once a week over a period of 8 weeks
  Interventions: Behavioral: Cognitive remediation

INTERVENTIONS:
Behavioral: D-MCT — Metacognitive Training for Depression (D-MCT), 8 sessions (60min); once a week over a period of 8 weeks. Metacognitive Training for depression (D-MCT) is a low-threshold, easy to administer group intervention. It aims at the reduction of depressive symptoms by changing cognitive biases; not only biases targeted in cognitive behavioral therapy but also those identified by basic research.
  Other Names: Metacognitive Training for Depression
  Arms: D-MCT Group
Behavioral: Cognitive remediation — A computerized cognitive remediation program that covers several cognitive domains, such as attention, visuomotor skills, and Memory. The difficulty level adapts automatically to the performance level of each patient. At the end of each session, the patient receives individual feedback on his or her performance; 8 sessions (60min), once a week over a period of 8 weeks
  Arms: Cognitive remediation

SUMMARY:
Aim of the current study is to investigate the acceptance and efficacy of Metacognitive Training for Depression (D-MCT) compared to cognitive remediation in outpatients with major depressive disorders in a randomized, controlled, assessor-blind, group trial.

DETAILED DESCRIPTION:
Evidence-based treatments for depression include pharmacological and psychological interventions. Within psychological interventions, cognitive behavioral therapy (CBT) is one of the most extensively researched evidence-based approaches for depression (Cuijpers, 2015). However, even if optimal treatment and access to services were available to all patients, the burden of depression would be reduced by only 30% (Andrews et al., 2004). Moreover, as depression represents the disorder with the highest drop-out rates during CBT treatment (36.4%) (Fernandez et al., 2015), and a relapse rate of 54% for treatment responders within the two years after treatment termination (Vittengl et al., 2007), it is pivotal to improve treatment for depression. It has been argued that this is less a question of developing novel psychological treatments as of determining how existing treatments may be improved (Cuijpers, 2015) and better disseminated to increase retention rates and to use the waiting phase to rise interest in therapy (Fernandez et al., 2015). Due to hopelessness and the discouraging character of the disorder, this poses a particular challenge.

To meet this aim, Metacognitive Training for Depression (D-MCT) has been developed as a low-threshold, highly standardized and yet easy to administer group concept for the treatment of depression. It is conceptualized as a variant of CBT that adopts a metacognitive perspective focusing on the modification of cognitive biases, and is compatible with a general CBT treatment approach. Use of standardized presentations reduces time needed for preparation and administration of the training; moreover, this "packaging" increases the accessibility of D-MCT to a wide range of health care providers, and encourages standardization across therapists. The training seeks to enable group members to recognize and correct the often automatic and unconscious thought patterns that accompany depression. To this end, it attempts to challenge cognitive biases through the use of creative and engaging exercises supported by a multimedia presentation (e.g., insight based on "aha" effects rather than psychoeducation) and to encourage patients to take a metacognitive perspective ("think about one's thinking"). The training is highly flexible with regard to depth and intensity. Patients do not need to (but may) discuss their own problems, and can still experience how cognitive biases work and influence one's mood in a playful atmosphere. The training is conceptualized as an open group: New patients can join the group in every session. Thus, the threshold for administration of and participation in this intervention is low.

The general structure of and exercises in D-MCT were inspired by Metacognitive Training for psychosis (Moritz et al., 2014); however, contents were modified upon to suit the specific problems of individuals with depression. Beside depressive thought patterns already targeted in CBT (e.g., overgeneralization, "mind reading"), a number of general cognitive biases, which have been identified by basic cognitive research, form the core of D-MCT (e.g., mood-congruent memory (Mathews and MacLeod, 2005)). Finally, as in Metacognitive Therapy (MCT) sensu Adrian Wells (Wells, 2011) dysfunctional coping strategies (i.e., thought suppression, rumination as problem-solving) are challenged. D-MCT thus blends established elements from CBT and MCT as well as newly developed and evidence-based exercises in one coherent metacognitive approach.

D-MCT was positively evaluated with regard to feasibility and acceptance in a non-randomized pilot study (Jelinek et al., 2013). Moreover, efficacy of D-MCT was suggested in a randomized controlled trail (RCT) in comparison to an active control intervention (Jelinek et al., 2016). In this trial patients with depressive disorder were completing a psychosomatic outpatient treatment program and were randomly assigned to either D-MCT or general health training. Severity of depression and cognitive biases were assessed at baseline (t0), post treatment (t1) and 6 months (t2) later by raters blind to diagnostic status. Intention-to-treat analyses demonstrated that at the end of treatment, as well as 6 months later, improvement in depression was significantly greater in the D-MCT relative to the health training group at medium effect sizes. A significantly greater number of patients in the D-MCT group were in remission at 6-month follow-up. Moreover, the decrease in cognitive biases and increase in psychological well-being/quality of life was larger in the D-MCT than the health training group over time. Patients' subjective appraisal of D-MCT was also positive (Jelinek et al., 2017).

Aim of the current study is to investigate the acceptance and efficacy of D-MCT in outpatients.The Hamilton Depression Rating Scale (HDRS, 17-item version) total score as well as the Quick Inventory of Depressive Symptomatology (QIDS) serve as primary outcome. Self-assessed depression, dysfunctional beliefs, self-esteem, quality of life, rumination, remission rate as well as neuropsychological functioning serve as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* age between 18 and 70 years
* diagnosis of a single Episode or recurrent Major depressive disorder (MDD) or dysthymia (verified by the MINI)

Exclusion Criteria:

* lifetime psychotic symptoms (i.e., hallucinations, delusions, or mania), suicidality (Suicidal Behaviors Questionnaire-Revised ≥ 7), intellectual disability (estimated IQ < 70) or dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology (QIDS) | eight months from baseline (t0) to 6-months follow up (t2)
  Primary outcome is change on the Quick Inventory of Depressive Symptomatology (QIDS) from baseline to follow-up (t0 - t2)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | [Time Frame: eight months from baseline (t0) to 6-months follow up (t2)]
  Change on the Hamilton Depression Rating Scale (HDRS, 17-item version) from baseline to follow-up (t0 - t2)
Self-assessed depression | [Time Frame: eight months from baseline (t0) to 6-months follow up (t2)]
  Change in self-assessed depression as measured by the Patient Health Questionnaire (PHQ-9) from baseline to follow-up (t0 to t2)
Quick Inventory of Depressive Symptomatology (QIDS) | from baseline (t0) to post intervention assessment at 8 weeks (t1) [time frame: 8 weeks]
  Change on the Quick Inventory of Depressive Symptomatology (QIDS) from baseline to post intervention assessment (t0 - t1)
Hamilton Depression Rating Scale | from baseline (t0) to post intervention assessment at 8 weeks (t1) [time frame: 8 weeks]
  Change on the Hamilton Depression Rating Scale from baseline to post intervention assessment (t0 - t1)
Patient Health Questionnaire (PHQ-9) | from baseline (t0) to post intervention assessment at 8 weeks (t1) [time frame: 8 weeks]
  Change on the Patient Health Questionnaire (PHQ-9) from baseline to post intervention assessment (t0 - t1)
Dysfunctional beliefs | eight months from baseline (t0) to 6-months follow up (t2
  Change in dysfunctional beliefs as measured by the Dysfunctional Attitude Scale (DAS) from baseline to follow-up (t0 to t2)
Quality of life | eight months from baseline (t0) to 6-months follow up (t2)
  Change in quality of life as measured by the World Health Organization Quality of Life Assessment (WHOQOL-BREF) from baseline to follow-up (t0 to t2)
Dysfunctional metacognitive beliefs | eight months from baseline (t0) to 6-months follow up (t2)
  Change in metacognitive beliefs as measured by the Metacognitions Questionnaire (MCQ-30) from baseline to follow-up (t0 to t2)
Rumination | eight months from baseline (t0) to 6-months follow up (t2)
  Rumination measured by the Ruminative Response Scale (RRS) from baseline to follow-up (t0 to t2)
Self-esteem | eight months from baseline (t0) to 6-months follow up (t2)
  Change in self-esteem as measured by the Rosenberg Self-Esteem Scale (RSE) from from baseline to follow-up (t0 to t2)
Remission rate | eight months from baseline (t0) to 6-months follow up (t2)
  Remission rate at T2 as measured by the Hamilton Depression Rating Scale (HDRS score ≤ 8)
Information processing | from baseline (t0) to post intervention assessment at 8 weeks (t1) [time frame: 8 weeks]
  Information processing as measured by the Trail-Making Test A (TMT-A) from baseline to post treatment assessment (t0 to t1)
Subjective appraisal of the training | each week (session data) [time frame: 8 weeks] and six months from post treatment assessment (t1) to 6 months follow up (t1 to t2) [time frame: 6 months]
  Subjective appraisal of the training after each session as well as at post treatment and follow up assessment (for questionnaire see Jelinek et al., 2017)
Executive functioning | from baseline (t0) to post intervention assessment at 8 weeks (t1) [time frame: 8 weeks]
  Executive functions as measured by the Trail-Making Test B (TMT-B) from baseline to post treatment assessment (t0 to t1)
Verbal memory | from baseline (t0) to post intervention assessment at 8 weeks (t1) [time frame: 8 weeks]
  Memory functioning as measured by Rivermead Behavioral Memory Test from baseline to post treatment assessment (t0 to t1)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Hagemann-Goebel, Dr., Principal Investigator — Asklepios Klinik Nord-Ochsenzoll
Locations (1):
- Asklepios Klinik Nord-Ochsenzoll, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moritz S, Veckenstedt R, Andreou C, Bohn F, Hottenrott B, Leighton L, Kother U, Woodward TS, Treszl A, Menon M, Schneider BC, Pfueller U, Roesch-Ely D. Sustained and "sleeper" effects of group metacognitive training for schizophrenia: a randomized clinical trial. JAMA Psychiatry. 2014 Oct;71(10):1103-11. doi: 10.1001/jamapsychiatry.2014.1038. PMID 25103718
- [Background] Jelinek L, Hauschildt M, Wittekind CE, Schneider BC, Kriston L, Moritz S. Efficacy of Metacognitive Training for Depression: A Randomized Controlled Trial. Psychother Psychosom. 2016;85(4):231-4. doi: 10.1159/000443699. Epub 2016 May 27. No abstract available. PMID 27230865
- [Background] Jelinek L, Otte C, Arlt S, & Hauschildt M. Denkverzerrungen erkennen und korrigieren: Eine Machbarkeitsstudie zum Metakognitiven Training bei Depressionen (D-MKT). [Identifying and correcting cognitive biases: A Pilot study on the Metacognitive Training for Depression (D-MCT)] Zeitschrift für Psychiatrie, Psychologie und Psychotherapie, 61, 247-254, 2013.
- [Background] Jelinek L, Moritz S, Hauschildt M. Patients' perspectives on treatment with Metacognitive Training for Depression (D-MCT): Results on acceptability. J Affect Disord. 2017 Oct 15;221:17-24. doi: 10.1016/j.jad.2017.06.003. Epub 2017 Jun 7. PMID 28628763
- [Background] Andrews G, Issakidis C, Sanderson K, Corry J, Lapsley H. Utilising survey data to inform public policy: comparison of the cost-effectiveness of treatment of ten mental disorders. Br J Psychiatry. 2004 Jun;184:526-33. doi: 10.1192/bjp.184.6.526. PMID 15172947
- [Background] Cuijpers P. Psychotherapies for adult depression: recent developments. Curr Opin Psychiatry. 2015 Jan;28(1):24-9. doi: 10.1097/YCO.0000000000000121. PMID 25415495
- [Background] Fernandez E, Salem D, Swift JK, Ramtahal N. Meta-analysis of dropout from cognitive behavioral therapy: Magnitude, timing, and moderators. J Consult Clin Psychol. 2015 Dec;83(6):1108-22. doi: 10.1037/ccp0000044. Epub 2015 Aug 24. PMID 26302248
- [Background] Mathews A, MacLeod C. Cognitive vulnerability to emotional disorders. Annu Rev Clin Psychol. 2005;1:167-95. doi: 10.1146/annurev.clinpsy.1.102803.143916. PMID 17716086
- [Background] Vittengl JR, Clark LA, Dunn TW, Jarrett RB. Reducing relapse and recurrence in unipolar depression: a comparative meta-analysis of cognitive-behavioral therapy's effects. J Consult Clin Psychol. 2007 Jun;75(3):475-88. doi: 10.1037/0022-006X.75.3.475. PMID 17563164
- [Background] Wells, A., 2011. Metacognitive Therapy for anxiety and depression. The Guilford Press, New York.